CLINICAL TRIAL: NCT00616499
Title: A Phase II Trial of Neoadjuvant Gefitinib Therapy Based on Mutation Study in Biopsy- Proven Stage IIIA N2 Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Gefitinib in Treating Patients With Stage IIIA Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582623; YONSEI-4-2006-0136; ZENECA-YONSEI-4-2006-0136
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-09

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Gefitinib; Neoadjuvant Therapy

INTERVENTIONS:
Drug: gefitinib
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving Gefitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response rate to gefitinib treatment as preoperative induction therapy in patients with biopsy-proven stage IIIA (pN2) non-squamous non-small cell lung cancer accompanied by epidermal growth factor receptor (EGFR) mutations.

Secondary

* To determine the complete resection rate in patients treated with this drug.
* To determine the overall survival rate in patients treated with this drug.
* To determine the disease-free survival rate in patients treated with this drug.
* To determine the pathologic complete response rate in patients treated with this drug.
* To determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once a day on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients with resectable disease may undergo surgery. Patients with unresectable disease may undergo surgery, chemotherapy, and/or radiotherapy.

After completion of study therapy, patients are followed for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven stage IIIA nonsquamous non-small cell lung cancer

  * pN2 disease proven by mediastinoscopy
* Meets any of the following criteria:

  * Never smoked
  * EGFR mutations (in exon 18, 19, or 21)*
  * FISH positive for EGFR* NOTE: *Irrespective of smoking history
* Presence of at least 1 unidimensionally measurable lesion on thoracic CT scan, according to RECIST
* Feasible to undergo pneumonectomy or lobectomy

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* FEV_1 ≥ 2.0 L in preoperative pulmonary function test
* Hemoglobin ≥ 9.0 g/dL
* WBC 4,000-12,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3.0 times ULN
* AST and ALT ≤ 3.0 times ULN
* Creatinine ≤ 1.5 times ULN
* Negative pregnancy test

Exclusion criteria:

* Severe complications or infections
* Pregnant or breast-feeding women
* Clinically significant heart disease
* Uncontrolled hepatitis, chronic liver disease, or diabetes mellitus
* Another active cancer except properly treated carcinoma in situ of the cervix or basal/squamous cell skin carcinoma

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy, chemotherapy, hormone therapy, or target therapy
* No other concurrent systemic anticancer therapies, including experimental drugs, chemotherapy, immunotherapy, or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Complete resection rate
Overall survival rate
Median disease-free survival
Complete pathological response rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Study Chair — Yonsei University
Locations (4):
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center at Yonsei University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center - University of Ulsan College of Medicine, Seoul